CLINICAL TRIAL: NCT03417245
Title: ATLAS-A/B: A Phase 3 Study to Evaluate the Efficacy and Safety of Fitusiran in Patients With Hemophilia A or B, Without Inhibitory Antibodies to Factor VIII or IX
Brief Title: A Study of Fitusiran (ALN-AT3SC) in Severe Hemophilia A and B Patients Without Inhibitors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC14769; ALN-AT3SC-004 (Other: Alnylam); 2016-001464-11 (EudraCT Number)
Record Dates: First submitted 2018-01-25; First posted 2018-01-31 (Actual); Results first posted 2022-02-04 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: RNAi therapeutic; Hemophilia A; Hemophilia B; Hemophilia A, Severe; Hemophilia B, Severe; Blood Coagulation Disorders, Inherited; Blood Coagulation Disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn; Genetic Diseases, X-Linked; Factor VIII; Factor IX; Coagulants; Fitusiran
MeSH Terms: conditions — Hemophilia A; Hemophilia B; Blood Coagulation Disorders, Inherited; Blood Coagulation Disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn; Genetic Diseases, X-Linked | interventions — fitusiran; prothrombin complex concentrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Factor On-demand (Experimental): Participants received on-demand factor concentrates (as needed, for episodic bleeding episodes, and not on a regular regimen intended to prevent spontaneous bleeding) per Investigator discretion for the treatment of breakthrough bleeding episodes from Day 1 up to a total of 9 months.
  Interventions: Drug: factor concentrates
- Fitusiran 80 mg Prophylaxis (Experimental): Participants received open-label fitusiran 80 milligram (mg) administered subcutaneously (SC) as prophylaxis once monthly from Day 1 up to a total of 9 months. Participants received on-demand factor concentrates (per investigator's discretion and within bleeding dosing guidelines) for the treatment of breakthrough bleeding episodes.
  Interventions: Drug: fitusiran; Drug: factor concentrates

INTERVENTIONS:
Drug: fitusiran — by SC injection
  Arms: Fitusiran 80 mg Prophylaxis
Drug: factor concentrates — by intravenous (IV) injection

SUMMARY:
Primary Objective:

-To evaluate the efficacy of fitusiran compared to on-demand treatment with factor concentrates, as determined by the frequency of bleeding episodes.

Secondary Objectives:

* To evaluate the efficacy of fitusiran compared to on-demand treatment with factor concentrates, as determined by:

  * The frequency of spontaneous bleeding episodes.
  * The frequency of joint bleeding episodes.
  * Health-related quality of life (HRQOL) in participants >=17 years of age.
* To determine the frequency of bleeding episodes during the onset period.
* To determine the safety and tolerability of fitusiran.

DETAILED DESCRIPTION:
The duration of treatment with fitusiran was 9 months. The estimated total time on study, inclusive of screening, was up to 11 months for all participants in the factor on-demand arm and for participants in the fitusiran arm who enrolled in the extension study (LTE15174). The estimated total time on the study was up to 17 months for participants in the fitusiran treatment arm who did not enroll in the extension study due to the requirement for up to an additional 6 months of follow-up monitoring for antithrombin levels.

Participants who completed the study will be eligible for an open-label extension study LTE15174 (NCT03754790).

ELIGIBILITY:
Inclusion Criteria:

* Males, >=12 years of age.
* Severe hemophilia A or B without inhibitors.

  * Severity confirmed by a central laboratory where FVIII level was less than (<) 1 percent (%) or Factor IX (FIX) level was less than or equal to (<=) 2% at Screening.
  * On-demand use of factor concentrate to manage bleeding episodes for at least the last 6 months prior to Screening, and meet each of the following criterion:

    * Nijmegen modified Bethesda assay inhibitor titer of <0.6 Bethesda units per milliliter (BU/mL) at Screening.
    * No use of Bypassing agents to treat bleeding episodes for at least the last 6 months prior to Screening.
    * No history of immune tolerance induction therapy within the last 3 years prior to Screening.
* A minimum of 6 bleeding episodes requiring factor concentrate treatment within the last 6 months prior to Screening.
* Willing and complied with the study requirements and to provide written informed consent and assent.

Exclusion Criteria:

* Known co-existing bleeding disorders other than hemophilia A or B, i.e., Von Willebrand's disease, additional factor deficiencies, or platelet disorders.
* Antithrombin (AT) activity <60% at Screening.
* Co-existing thrombophilic disorder.
* Clinically significant liver disease.
* Active hepatitis C virus infection.
* HIV positive with a cluster of differentiation-4 count of <200 cells/microliter.
* History of arterial or venous thromboembolism.
* Inadequate renal function.
* History of multiple drug allergies or history of allergic reaction to an oligonucleotide or N-Acetylgalactosamine (GalNAc).
* History of intolerance to SC injection(s).
* Any other conditions or comorbidities that would make the participant unsuitable for enrollment or could interfere with participation in or completion of the study, per Investigator judgment.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, MD, Study Director — Sanofi
Locations (64):
- United States (8):
  - Investigational Site Number 0140, Little Rock, Arkansas
  - Investigational Site Number 128, Gainesville, Florida
  - Investigational Site Number 103, Tampa, Florida
  - Investigational Site Number 102, Chicago, Illinois
  - Investigational Site Number 119, New Orleans, Louisiana
  - Investigational Site Number 125, Ann Arbor, Michigan
  - Investigational Site Number 111, Las Vegas, Nevada
  - Investigational Site Number 110, Akron, Ohio
- Australia (3):
  - Investigational Site Number 6101, Camperdown
  - Investigational Site Number 6103, Murdoch
  - Investigational Site Number 6104, Prahran
- China (5):
  - Investigational Site Number 8604, Beijing
  - Investigational Site Number 8602, Guangzhou
  - Investigational Site Number 8605, Hangzhou
  - Investigational Site Number 8603, Shanghai
  - Investigational Site Number 8601, Tianjin
- Investigational Site Number 4501, Copenhagen, Denmark
- France (3):
  - Investigational Site Number 3303, Lyon
  - Investigational Site Number 3305, Paris
  - Investigational Site Number 3301, Rouen
- Germany (3):
  - Investigational Site Number 4904, Berlin
  - Investigational Site Number 4905, Frankfurt am Main
  - Investigational Site Number 4906, Leipzig
- Investigational Site Number 3602, Budapest, Hungary
- India (8):
  - Investigational Site Number 9102, Bangalore
  - Investigational Site Number 9104, Jaipur
  - Investigational Site Number 9106, Lucknow
  - Investigational Site Number 9109, Mumbai
  - Investigational Site Number 9108, Mumbai
  - Investigational Site Number 9111, Mumbai
  - Investigational Site Number 9103, Pune
  - Investigational Site Number 9105, Vellore
- Investigational Site Number 9701, Ramat Gan, Israel
- Investigational Site Number 3904, Padua, Italy
- Japan (2):
  - Investigational Site Number 8105, Isehara
  - Investigational Site Number 8104, Saitama
- Malaysia (3):
  - Investigational Site Number 6004, Ampang
  - Investigational Site Number 6002, Johor Bahru
  - Investigational Site Number 6003, Kota Kinabalu
- South Africa (2):
  - Investigational Site Number 2701, Parktown
  - Investigational Site Number 2702, Port Elizabeth
- South Korea (3):
  - Investigational Site Number 8201, Busan
  - Investigational Site Number 8202, Daejeon
  - Investigational Site Number 8204, Seoul
- Investigational Site Number 3402, Madrid, Spain
- Taiwan (5):
  - Investigational Site Number 8807, Taichung
  - Investigational Site Number 8805, Taichung
  - Investigational Site Number 8804, Taipei
  - Investigational Site Number 8801, Taipei
  - Investigational Site Number 8808, Taoyuan District
- Turkey (Türkiye) (7):
  - Investigational Site Number 9002, Adana
  - Investigational Site Number 9004, Antalya
  - Investigational Site Number 9008, Gaziantep
  - Investigational Site Number 9005, Istanbul
  - Investigational Site Number 9003, Izmir
  - Investigational Site Number 9009, Kayseri
  - Investigational Site Number 9006, Samsun
- Ukraine (4):
  - Investigational Site Number 8001, Kyiv
  - Investigational Site Number 8003, Kyiv
  - Investigational Site Number 8002, Lviv
  - Investigational Site Number 8005, Mykolaiv
- United Kingdom (3):
  - Investigational Site Number 4402, Glasgow
  - Investigational Site Number 4407, London
  - Investigational Site Number 4401, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Srivastava A, Rangarajan S, Kavakli K, Klamroth R, Kenet G, Khoo L, You CW, Xu W, Malan N, Frenzel L, Bagot CN, Stasyshyn O, Chang CY, Poloskey S, Qiu Z, Andersson S, Mei B, Pipe SW. Fitusiran prophylaxis in people with severe haemophilia A or haemophilia B without inhibitors (ATLAS-A/B): a multicentre, open-label, randomised, phase 3 trial. Lancet Haematol. 2023 May;10(5):e322-e332. doi: 10.1016/S2352-3026(23)00037-6. Epub 2023 Mar 29. PMID 37003278
- [Derived] Del Pozo Martin Y. 2021 ASH annual meeting. Lancet Haematol. 2022 Feb;9(2):e92-e93. doi: 10.1016/S2352-3026(21)00384-7. Epub 2021 Dec 16. No abstract available. PMID 34922648

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 64 centers in 19 countries. A total of 177 participants were screened between 1 March 2018 to 22 May 2020, of which 57 participants were screen failure. Screen failures were mainly due to presence of a co-existing thrombophilic disorder. In total, 120 participants were enrolled in the study.
Pre-assignment Details: 120 participants were randomized in 2:1 ratio to fitusiran prophylaxis and on-demand arms by interactive response system; stratified by the number of bleeding episodes in the 6 months prior to Screening (less than or equal to [<=10] versus greater than [>]10) and by hemophilia type (hemophilia A or B).
Period: Overall Study
Arm/Group | Factor On-demand | Fitusiran 80 mg Prophylaxis
Started | 40 | 80
Treated | 40 | 79
Completed | 37 | 79
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on intent-to-treat (ITT) population which included all randomized participants analyzed according to the randomized arm.
Arm/Group | Factor On-demand | Fitusiran 80 mg Prophylaxis | Total Title
Number analyzed (Participants) | 40 | 80 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (13.6) | 33.9 (14.6) | 33.8 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 40 | 80 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 28 | 43 | 71
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 12 | 33 | 45
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Estimated Annualized Bleeding Rate (ABR) for Treated Bleeds During the Efficacy Period
Description: ABR for a participant during efficacy period (EP) was defined as annualized number of bleeding episodes during EP annualized to a 1-year interval of time. Treated Bleeding episode: any occurrence of hemorrhage that required administration of by-passing agents (BPA) or factor. It started from first sign of a bleed and ended no more than 72 hours after last treatment for bleed, within which any symptoms of bleeding at same location or injections less than or equal to (<=) 72 hours apart were considered the same bleeding episode. EP was defined as time duration starting from Day 29 when antithrombin (AT) lowering capacity of fitusiran had achieved therapeutic target range to the earliest of Day 246 or last day of bleeding follow up (maximum duration of EP: from Day 29 to Day 246). This outcome measure (OM) presents estimated results (i.e., results received by applying negative binomial [NB] regression model on data collected during EP).
Time Frame: From Day 29 up to Day 246 or up to the last day of bleeding follow up (any day up to Day 246), whichever was the earliest
Population: Analysis was performed on ITT population. Here, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | Factor On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 40 | 79
episodes per participant per year | 30.991 [21.114 to 45.487] | 3.133 [2.269 to 4.326]
Statistical Analysis 1: Comparison: Factor On-demand vs Fitusiran 80 mg Prophylaxis; Test type: Superiority; p < 0.0001, Negative binomial regression mode — P-value derived from NB regression model during EP, with treatment arm, number of bleeds in 6 months prior to study (<=10, >10) and hemophilia type (A vs B) as fixed effects. Significance threshold was at 0.05; ABR ratio = 0.101, 95% CI 2-sided [0.064 to 0.159]

2. Primary Outcome: Observed Annualized Bleeding Rate (ABR) for Treated Bleeds During the Efficacy Period
Description: ABR for a participant during EP was defined as annualized number of bleeding episodes during EP annualized to a 1-year interval of time. ABR= number of bleeding episodes during EP divided by total number of days during EP*365.25. A bleeding episode was defined as any occurrence of hemorrhage that required administration of BPA or factor. It started from the first sign of a bleed and ended no more than 72 hours after the last treatment for the bleed, within which any symptoms of bleeding at the same location or injections <=72 hours apart were considered the same bleeding episode. EP was defined as time duration starting from Day 29 when the AT lowering capacity of fitusiran had achieved therapeutic target range to the earliest of Day 246 or the last day of bleeding follow up (maximum duration of EP: from Day 29 to Day 246). This OM presents observed results (i.e., descriptive statistics values based on the data collected during EP).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Arm/Group | Factor On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 40 | 79
episodes per participant per year | 21.8 [8.4 to 41.0] | 0.0 [0.0 to 3.4]

3. Secondary Outcome: Estimated Annualized Bleeding Rate (ABR) for Treated Bleeds During the Treatment Period
Description: ABR for a participant during treatment period (TP) was defined as annualized number of bleeding episodes during TP annualized to a 1-year interval of time. Bleeding episode: any occurrence of hemorrhage that required administration of BPA or factor. It started from first sign of a bleed and ended no more than 72 hours after last treatment for bleed, within which any symptoms of bleeding at same location or injections <=72 hours apart were considered the same bleeding episode. TP was sum of onset period (first 28 days after first dose of fitusiran) and EP (starting on Day 29 when AT lowering capacity of fitusiran had achieved therapeutic target range to earliest of Day 246 or last day of bleeding follow up (maximum duration of TP: from Day 1 to Day 246). This OM presents estimated results (i.e., results received by applying NB regression model on data collected during TP).
Time Frame: From Day 1 up to Day 246 or up to the last day of bleeding follow up (any day up to Day 246), whichever was the earliest
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | Factor On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 40 | 79
episodes per participant per year | 31.444 [22.995 to 42.999] | 4.092 [3.143 to 5.328]
Statistical Analysis 1: Comparison: Factor On-demand vs Fitusiran 80 mg Prophylaxis; Test type: Superiority; p < 0.0001, Negative binomial regression model — P-value derived from NB regression model during TP, with treatment arm, number of bleeds in 6 months prior to study (<=10, >10) and hemophilia type (A vs B) as fixed effects. Significance threshold was at 0.05; ABR ratio = 0.130, 95% CI 2-sided [0.090 to 0.188]

4. Secondary Outcome: Observed Annualized Bleeding Rate (ABR) for Treated Bleeds During the Treatment Period
Description: ABR for a participant during TP was defined as annualized number of bleeding episodes during TP annualized to a 1- year interval of time. ABR= number of bleeding episodes during TP divided by total number of days during TP*365.25. Bleeding episode: any occurrence of hemorrhage that required administration of BPA or factor. It started from the first sign of a bleed and ended no more than 72 hours after last treatment for bleed, within which any symptoms of bleeding at the same location or injections <=72 hours apart were considered the same bleeding episode. TP was sum of onset period (first 28 days after the first dose of fitusiran) and EP (starting on Day 29 when AT lowering capacity of fitusiran had achieved therapeutic target range to the earliest of Day 246 or the last day of bleeding follow up (maximum duration of TP: from Day 1 to Day 246). This OM presents observed results (i.e., descriptive statistics values based on data collected during TP).
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Arm/Group | Factor On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 40 | 79
episodes per participant per year | 25.2 [11.9 to 43.8] | 1.8 [0.0 to 4.5]

5. Secondary Outcome: Estimated Annualized Spontaneous Bleeding Rate for Treated Bleeds During the Efficacy Period
Description: Annualized spontaneous bleeding rate for a participant during EP was defined as annualized number of spontaneous bleeding episodes during EP annualized to a 1-year interval of time. Spontaneous bleeding episode was bleeding event that occurred for no apparent or known reason, particularly into joints, muscles, and soft tissues. It started from first sign of a bleed and ended no more than 72 hours after last treatment for the bleed, within which any symptoms of bleeding at the same location or injections <=72 hours apart were considered the same bleeding episode. EP was defined as time duration starting from Day 29 when AT lowering capacity of fitusiran had achieved therapeutic target range to the earliest of Day 246 or last day of bleeding follow up (maximum duration of EP: from Day 29 to Day 246). This OM presents estimated results (i.e., results received by applying NB regression model on data collected during EP).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | Factor On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 40 | 79
episodes per participant per year | 22.036 [14.159 to 34.295] | 1.825 [1.237 to 2.692]
Statistical Analysis 1: Comparison: Factor On-demand vs Fitusiran 80 mg Prophylaxis; Test type: Superiority; p < 0.0001, Negative binomial regression model — [p-value comment as in outcome 1, analysis 1]; ABR ratio = 0.083, 95% CI 2-sided [0.049 to 0.141]

6. Secondary Outcome: Observed Annualized Spontaneous Bleeding Rate for Treated Bleeds During the Efficacy Period
Description: ABR for participant during EP was defined as annualized number of spontaneous bleeding episodes during EP annualized to a 1-year interval of time. ABR=number of treated spontaneous bleeding episodes during EP divided by total number of days during EP*365.25. Spontaneous bleeding episode was bleeding event that occurred for no apparent or known reason, into joints, muscles, and soft tissues. It started from the first sign of a bleed and ended no more than 72 hours after the last treatment for the bleed, within which any symptoms of bleeding at the same location or injections <=72 hours apart were considered the same bleeding episode. EP: time duration starting from Day 29 when the AT lowering capacity of fitusiran had achieved therapeutic target range to earliest of Day 246 or the last day of bleeding follow up (maximum duration of EP: from Day 29 to Day 246).This OM presents observed results (i.e., descriptive statistics values based on data collected during EP).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Arm/Group | Factor On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 40 | 79
episodes per participant per year | 16.1 [3.4 to 27.6] | 0.0 [0.0 to 1.7]

7. Secondary Outcome: Estimated Annualized Joint Bleeding Rate for Treated Bleeds During the Efficacy Period
Description: Annualized joint bleeding rate for a participant during EP was defined as annualized number of bleeding episodes during EP annualized to a 1-year interval of time. Joint bleeding episode was characterized by an unusual sensation in the joint ("aura") in combination with 1) increasing swelling or warmth over the skin, joint, 2) increasing pain, or 3) progressive loss of range of motion or difficulty in using the limb as compared with Baseline. It started from first sign of a bleed and ended no more than 72 hours after last treatment for the bleed. EP was defined as time duration starting from Day 29 when the AT lowering capacity of fitusiran had achieved therapeutic target range to the earliest of Day 246 or the last day of bleeding follow up (maximum duration of EP: from Day 29 to Day 246). This OM presents estimated results (i.e., results received by applying NB regression model on data collected during EP).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | Factor On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 40 | 79
episodes per participant per year | 23.413 [15.363 to 35.680] | 2.282 [1.594 to 3.268]
Statistical Analysis 1: Comparison: Factor On-demand vs Fitusiran 80 mg Prophylaxis; Test type: Superiority; p < 0.0001, Negative binomial regression model — [p-value comment as in outcome 1, analysis 1]; ABR ratio = 0.097, 95% CI 2-sided [0.059 to 0.161]

8. Secondary Outcome: Observed Annualized Joint Bleeding Rate for Treated Bleeds During the Efficacy Period
Description: Annualized joint bleeding rate for participant during EP was defined as annualized number of joint bleeding episodes during EP annualized to 1-year interval of time. ABR= number of treated joint bleeding episodes during EP divided by total number of days during EP*365.25. A joint bleeding episode was characterized by an unusual sensation in joint ("aura") in combination with 1) increasing swelling or warmth over skin, joint, 2) increasing pain, or 3) progressive loss of range of motion or difficulty in using limb as compared with Baseline. It started from first sign of a bleed and ended no more than 72 hours after the last treatment for the bleed. EP: time duration starting from Day 29 when the AT lowering capacity of fitusiran had achieved therapeutic target range to the earliest of Day 246 or last day of bleeding follow up (maximum duration of EP: from Day 29 to Day 246). This OM presents observed results (i.e., descriptive statistics values based on data collected during EP).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Arm/Group | Factor On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 40 | 79
episodes per participant per year | 15.9 [4.2 to 33.5] | 0.0 [0.0 to 3.4]

9. Secondary Outcome: Health-related Quality of Life (HRQOL): Change From Baseline in Haemophilia Quality of Life Questionnaire for Adults (Haem-A-QOL) Physical Health Score at Month 9
Description: Haem-A-QoL: participant-reported questionnaire designed for adult participants (>=17 years of age) with hemophilia; and consisted of 46 items comprising 10 domains (physical health, feelings, view of yourself, sports and leisure, work and school, dealing with hemophilia, treatment, future, family planning, partnership and sexuality). Scoring for each item was based on a 5-point Likert scale (1= never, 2= rarely, 3= sometimes, 4= often, and 5=all the time), and higher scores represented greater impairment. Change from baseline in physical health domain score was reported in this outcome measure. Raw score for physical health domain were transformed to a scale ranged from 0 (better health outcome) to 100 (worst health outcome), where lower scores denoted better physical health.
Time Frame: Baseline (Day 1), Month 9
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Factor On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 34 | 69
scores on a scale | -3.32 [-9.67 to 3.04] | -23.07 [-28.00 to -18.14]
Statistical Analysis 1: Comparison: Factor On-demand vs Fitusiran 80 mg Prophylaxis; Test type: Superiority; p < 0.0001, ANCOVA — Analysis of Covariance (ANCOVA) model included treatment arm, number of bleeds in 6 months prior to study (<=10,>10) and hemophilia type (A vs B) as fixed effects, Baseline score as covariate. Significance threshold was at 0.05; Least Square (LS) Mean difference = -19.75, 95% CI 2-sided [-27.00 to -12.50]

10. Secondary Outcome: Health-related Quality of Life (HRQOL): Change From Baseline in Haem-A-QOL Total Score at Month 9
Description: Haem-A-QoL: participant-reported questionnaire designed for adult participants (>=17 years of age) with hemophilia; and consisted of 46 items comprising 10 domains (physical health, feelings, view of yourself, sports and leisure, work and school, dealing with hemophilia, treatment, future, family planning, partnership and sexuality). Scoring for each item was based on a 5-point Likert scale (1= never, 2= rarely, 3= sometimes, 4= often, and 5=all the time), and higher scores represent greater impairment. Raw score for each domain were transformed to a scale ranged between 0 and 100, where lower scores denoted better health. Haem-A-QoL total score was average of all domain scores and ranged from 0 (better health outcome) to 100 (worst health outcome), where lower scores denoted better physical health.
Time Frame: Baseline (Day 1), Month 9
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Factor On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 34 | 69
scores on a scale | -2.62 [-6.27 to 1.03] | -9.68 [-12.51 to -6.86]
Statistical Analysis 1: Comparison: Factor On-demand vs Fitusiran 80 mg Prophylaxis; Test type: Superiority; p = 0.0011, ANCOVA — ANCOVA model included treatment arm, number of bleeds in 6 months prior to study (<=10,>10) and hemophilia type (A vs B) as fixed effects, Baseline score as covariate. Significance threshold was at 0.05; LS Mean difference = -7.07, 95% CI 2-sided [-11.23 to -2.90]

11. Secondary Outcome: Estimated Annualized Bleeding Rate (ABR) for Treated Bleeds During the Onset Period
Description: ABR was annualized number of bleeding episodes during onset period per participant annualized to a 1-year interval of time. A treated bleeding episode was defined as any occurrence of hemorrhage that required administration of BPA or factor. It started from the first sign of a bleed and ended no more than 72 hours after the last treatment for the bleed, within which any symptoms of bleeding at the same location or injections <=72 hours apart were considered the same bleeding episode. The onset period was defined as time interval from Day 1 to the earlier of Day 28 or the last day of bleeding follow up. This OM presents estimated results (i.e., results received by applying NB regression model on data collected during onset period).
Time Frame: From Day 1 up to Day 28 or up to the last day of bleeding follow up (any day up to Day 28), whichever was the earliest
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | Factor On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 40 | 79
episodes per participant per year | 33.389 [25.619 to 43.517] | 10.805 [8.143 to 14.337]

12. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug which did not necessarily have a causal relationship with the treatment. Treatment-emergent AEs were defined as any AE with onset date after first dose of fitusiran in the fitusiran prophylaxis arm or after Day 1 visit in the factor on-demand arm. A serious AE (SAE) was defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability or incapacity, was a congenital anomaly or birth defect, or was a medically important event.
Time Frame: From Baseline (Day 1) up to 15 months (i.e., 9 months treatment period + 6-month follow-up)
Population: Analysis was performed on safety analysis set that included all participants who received at least 1 dose of study drug or were randomized to on-demand arm, analyzed according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Factor On-demand | Fitusiran 80 mg Prophylaxis
Number analyzed (Participants) | 40 | 79
Participants
  Any TEAE | 18 | 62
  Any TESAE | 5 | 5

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1) up to 15 months (i.e., 9 months treatment period + 6-month follow-up).
Description: Treatment-emergent AE were defined as any AE with onset date after first dose of fitusiran in the fitusiran prophylaxis arm or after Day 1 visit in the factor on-demand arm. Analysis was performed on safety analysis set.
Arm/Group | Factor On-demand | Fitusiran 80 mg Prophylaxis
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/79
Serious Adverse Events (participants affected / at risk) | 5/40 | 5/79
Other Adverse Events (participants affected / at risk) | 8/40 | 45/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Factor On-demand (N=40) | Fitusiran 80 mg Prophylaxis (N=79)
Epidural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Factor On-demand (N=40) | Fitusiran 80 mg Prophylaxis (N=79)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 18 (20)
Aspartate Aminotransferase Increased (Investigations) | 2 (2) | 6 (7)
Blood Bilirubin Increased (Investigations) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 5 (6)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 6 (6)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 4 (5)
Gastritis (Gastrointestinal disorders) | 1 (1) | 5 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6)
Nasopharyngitis (Infections and infestations) | 3 (3) | 7 (7)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 9 (9)
Hypertension (Vascular disorders) | 4 (4) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT03417245/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/45/NCT03417245/SAP_001.pdf